CLINICAL TRIAL: NCT01830296
Title: COADMINISTRATION OF INTRAVENOUS REMIFENTANIL AND MORPHINE FOR POSTTHORACOTOMY PAIN; COMPARISON WITH IV MORPHINE ALONE
Brief Title: Intravenous Remifentanil Plus Morphine or Morphine Alone for Postthoracotomy Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Hakki Unlugenc, Prof Dr., Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MDHTRKTN13
Record Dates: First submitted 2013-03-27; First posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Pain
Keywords: Postthoracotomy pain,; patient controlled analgesia,; remifentanil and; morphine.
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanil+Morphine (Active Comparator): Morphine(M) Remifentanil+Morphine(MR)
  Interventions: Drug: Remifentanil+morphine
- IV morphine PCA (Active Comparator): IV remifentanil+morphine PCA
  Interventions: Drug: Remifentanil+morphine

INTERVENTIONS:
Drug: Remifentanil+morphine — Morphine, Remifentanil+Morphine
  Other Names: Morphine Group (M); Remifentanil+Morphine Group (MR)

SUMMARY:
Background; Post-thoracotomy pain remains a major problem. This double-blind, randomized study tested the effects of coadministration of patient controlled remifentanil+morphine combination on postthoracotomy pain, analgesic consumption and side effects compared with morphine PCA alone

DETAILED DESCRIPTION:
Methods; Sixty patients were allocated randomly to receive an intravenous patient-controlled analgesia with morphine alone (M), or morphine plus remifentanil (MR), in a double-blind manner. Postoperatively patients were allowed to use bolus doses of morphine (0.2 mg kg-1) or morphine (0.2 mg kg-1) plus remifentanil (0.2 µg kg-1) mixture every 10 min without a background infusion. Pain, discomfort, sedation scores, total and bolus patient-controlled morphine consumption, rescue analgesic requirement and side-effects were recorded for up to 24 h after the start of patient-controlled analgesia.

ELIGIBILITY:
Inclusion Criteria:

* 60 ASA physical status I-III patients, between the ages of 18 and 59 years, scheduled for elective thoracotomy surgery with general anaesthesia were included in this study

Exclusion Criteria:

* severe hepatorenal disease history, sensitivity or contraindication to morphine and remifentanil, chronic pain (defined as regular use of opioid analgesics for > 3 months), drug or alcohol abuse and contraindication to administration of PCA

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
COADMINISTRATION OF INTRAVENOUS REMIFENTANIL AND MORPHINE FOR POSTTHORACOTOMY PAIN; COMPARISON WITH IV MORPHINE ALONE | Two years
  As aim of this study was to evaluate the effects of remifentanil addition to morphine for i.v. PCA on analgesic consumption, the primary endpoint was defined as morphine consumption at 24 hour.

CONTACTS AND LOCATIONS:
Overall Officials: Mediha Turktan, Assist Prof, Study Director — Cukurova University, Department of Anaesthesiology
Locations (1):
- Hakkı Unlugenc, Adana, Turkey (Türkiye)